CLINICAL TRIAL: NCT02107859
Title: An Open-Label Safety and Efficacy Study for Patients With Nonsense Mutation Cystic Fibrosis Previously Treated With Ataluren (PTC124)
Brief Title: Study of Ataluren (PTC124) in Cystic Fibrosis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on the results of study PTC124-GD-021-CF (NCT02139306), clinical development of ataluren in cystic fibrosis was discontinued and this study was closed.
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC124-GD-023-CF; 2013-005449-35 (EudraCT Number)
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Results first posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Nonsense mutation; Premature stop codon; PTC124; Ataluren
MeSH Terms: conditions — Cystic Fibrosis | interventions — ataluren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ataluren (Experimental): Participants will receive ataluren suspension orally 3 times a day (TID), 10 milligrams/kilogram (mg/kg) at morning, 10 mg/kg at midday, and 20 mg/kg at evening (total daily dose 40 mg/kg) for 192 weeks.
  Interventions: Drug: Ataluren

INTERVENTIONS:
Drug: Ataluren — Ataluren will be administered per dose and schedule specified in the arm.
  Other Names: PTC124

SUMMARY:
The primary objective of this study is to determine the long-term safety and tolerability of ataluren in participants with nonsense mutation cystic fibrosis (nmCF) who completed participation in the double-blind study PTC124-GD-009-CF (NCT00803205), as assessed by adverse events and laboratory abnormalities. The secondary objective of this study includes the assessment of the efficacy of ataluren, as measured by forced expiratory volume in 1 second (FEV1) and pulmonary exacerbation rate, and other safety parameters (for example, 12-lead electrocardiogram [ECG] measurements, vital signs).

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to provide written informed consent (parental/guardian consent and participant assent if less than [<] 18 years of age).
* Evidence of completed participation in the double-blind study, PTC124-GD-009-CF (Study 009).
* Body weight greater than or equal to (≥) 16 kilograms (kg).
* Performance of a valid, reproducible spirometry test using the study-specific spirometer during the screening period.
* Confirmed laboratory values within the central laboratory ranges at screening.
* In male and female participants who are sexually active, willingness to abstain from sexual intercourse or employ a barrier or medical method of contraception during the study drug administration and 60-day follow-up period.
* Willingness and ability to comply with all study procedures and assessments, including scheduled visits, drug administration plan, laboratory tests, and study restrictions.

Key Exclusion Criteria:

* Chronic use of systemic tobramycin within 4 weeks prior to screening.
* Evidence of pulmonary exacerbation or acute upper or lower respiratory tract infection (including viral illnesses) within 3 weeks prior to screening or between screening and randomization.
* Any change (initiation, change in type of drug, dose modification, schedule modification, interruption, discontinuation, or re-initiation) in a chronic treatment/prophylaxis regimen for CF or for CF-related conditions within 4 weeks prior to screening and randomization.
* Known hypersensitivity to any of the ingredients or excipients of the study drug.
* Exposure to another investigational drug within 4 weeks prior to screening.
* Treatment with intravenous antibiotics within 3 weeks prior to screening.
* History of solid organ or hematological transplantation.
* Ongoing immunosuppressive therapy (other than corticosteroids).
* Positive hepatitis B surface antigen, hepatitis C antibody test or human immunodeficiency virus (HIV) test.
* Known portal hypertension.
* Pregnancy or breast-feeding.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-05-23 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph McIntosh, MD, Study Director — PTC Therapeutics, Inc.
Locations (17):
- United States (7):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Miller Children's Hospital Long Beach, Long Beach, California
  - Denver Children's Hospital, Aurora, Colorado
  - Children's Hospital Chicago, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - Beth Israel Medical Center, New York, New York
  - Rainbow Babies & Children's Hospital, Cleveland, Ohio
- Belgium (3):
  - Hôpital Universitaire des Enfants Reine Fabiola, Brussels
  - University Hospital Brussels, Brussels
  - University Hospital Leuven, Leuven
- France (2):
  - Hôpital Necker - Enfants Malades, Paris
  - Hôpital des Enfants, Toulouse
- Hadassah University Hospital - Mount Scopus, Jerusalem, Israel
- Italy (2):
  - Università La Sapienza, Roma
  - Azienda Ospedaliera di Verona, Verona
- Hospital Universitario La Paz, Madrid, Spain
- Karolinska University Hospital, Huddinge, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aslam AA, Sinha IP, Southern KW. Ataluren and similar compounds (specific therapies for premature termination codon class I mutations) for cystic fibrosis. Cochrane Database Syst Rev. 2023 Mar 3;3(3):CD012040. doi: 10.1002/14651858.CD012040.pub3. PMID 36866921
- See also: PTC Therapeutics, Inc. website — http://www.ptcbio.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with nonsense mutation cystic fibrosis (nmCF) who had completed the double-blind study PTC124-GD-009-CF (NCT00803205) were enrolled and treated in this open-label extension study.
Pre-assignment Details: On 2 March 2017, it was announced that the Phase 3 double-blind study PTC124-GD-021-CF (NCT02139306) did not achieve its primary or secondary endpoints. Based on these results, clinical development of ataluren in cystic fibrosis was discontinued and this ongoing open-label extension study was closed.
Groups:
- Ataluren: Participants received ataluren suspension orally 3 times a day (TID), 10 milligrams/kilogram (mg/kg) at morning, 10 mg/kg at midday, and 20 mg/kg at evening (total daily dose 40 mg/kg) for 192 weeks.
Period: Overall Study
Arm/Group | Ataluren
Started | 61
As-treated Population (Received at .least 1 dose of study drug) | 61
Intent-to-treat (ITT) Population (All participants who had at least 1 post-baseline efficacy assessment.) | 60
Completed | 0
Not Completed | 61
Not completed — Withdrawal by Subject | 14
Not completed — Adverse Event | 3
Not completed — Study closure | 41
Not completed — Other than specified | 3

BASELINE CHARACTERISTICS:
Population: As-treated population included all participants who received at least 1 dose of ataluren.
Groups:
- Ataluren: Participants received ataluren suspension orally TID, 10 mg/kg at morning, 10 mg/kg at midday, and 20 mg/kg at evening (total daily dose 40 mg/kg) for 192 weeks.
Arm/Group | Ataluren
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White-White/Caucasian | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: AE: any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Severity of an AE was classified as: mild (does not interfere with usual function), moderate (interferes to some extent with usual function), severe (interferes significantly with usual function), life threatening (results in potential threat to life), and fatal AEs. Drug-related AEs: AEs with a possible or probable relationship to study drug. Serious AEs: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention. TEAE: AE that occurred or worsened from first dose of study drug to 4 weeks after last dose of study drug. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline (Day 1) up to end of study (Week 196)
Population: As-treated population included all participants who received at least 1 dose of ataluren.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren
Number analyzed (Participants) | 61
Participants
  Any TEAEs | 61
  Mild AEs | 4
  Moderate AEs | 26
  Severe AEs | 30
  Life-threatening AEs | 0
  Fatal AEs | 1
  AEs unrelated to ataluren | 35
  AEs unlikely related to ataluren | 12
  AEs possible related to ataluren | 13
  AEs probable related to ataluren | 1
  Serious TEAEs | 36

2. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Laboratory parameters tests included hematology, biochemistry assay (hepatic, renal, and serum electrolyte values), adrenal assays, and urinalysis. Clinical significance was defined as per investigator's judgement.
Time Frame: Baseline (Day 1) up to end of study (Week 196)
Population: As-treated population included all participants who received at least 1 dose of ataluren.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren
Number analyzed (Participants) | 61
Participants | 0

3. Secondary Outcome: Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) at the End of Treatment (Week 192), as Assessed by Spirometry
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Percent of predicted FEV1 = (observed value)/(predicted value) * 100%. Change from baseline in percent predicted FEV1 at the end of treatment was reported.
Time Frame: Baseline, Week 192
Population: ITT population included all participants who had at least 1 post-baseline efficacy assessment. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure. 'Number analyzed' signifies participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Ataluren
Number analyzed (Participants) | 59
percentage of predicted FEV1
  Baseline | 56.203 (17.2964)
  Change at Week 192: number analyzed (Participants) | 7
  Change at Week 192 | -1.214 (3.6384)

4. Secondary Outcome: Percentage of Participants With Pulmonary Exacerbation, As Assessed by Modified Fuchs Criteria
Description: The modified Fuchs' criteria defined exacerbation as the presence of at least 4 of the following 12 Fuchs' signs and symptoms without the requirement for treatment with antibiotics: change in sputum; new or increased hemoptysis; increased cough; increased dyspnea; fatigue; temperature greater than (>) 38 degrees celsius (°C); anorexia; sinus pain; change in sinus discharge; change in physical examination of the chest; decrease in pulmonary function by 10 percent or more from a previously recorded value; or radiographic changes indicative of pulmonary function.
Time Frame: Baseline up to Week 192
Population: ITT population included all participants who had at least 1 post-baseline efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Ataluren
Number analyzed (Participants) | 60
percentage of participants | 68.3

5. Secondary Outcome: Percentage of Participants With Pulmonary Exacerbation, As Assessed by Expanded Fuchs' Criteria
Description: The expanded Fuchs' criteria defined exacerbation as the presence of at least 4 of the following 12 Fuchs' signs and symptoms requiring any form of antibiotic treatment (inhaled, oral, or intravenous): change in sputum; new or increased hemoptysis; increased cough; increased dyspnea; fatigue; temperature >38°C; anorexia; sinus pain; change in sinus discharge; change in physical examination of the chest; decrease in pulmonary function by 10 percent or more from a previously recorded value; or radiographic changes indicative of pulmonary function.
Time Frame: Baseline up to Week 192
Population: ITT population included all participants who had at least 1 post-baseline efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Ataluren
Number analyzed (Participants) | 60
percentage of participants | 68.3

6. Secondary Outcome: Percentage of Participants With Pulmonary Exacerbation, As Assessed by Classic Fuchs' Criteria
Description: The Classic Fuchs' criteria defined exacerbation as the presence of at least 4 of the following 12 Fuchs' signs and symptoms requiring treatment with parenteral antibiotics: change in sputum; new or increased hemoptysis; increased cough; increased dyspnea; fatigue; temperature >38°C; anorexia; sinus pain; change in sinus discharge; change in physical examination of the chest; decrease in pulmonary function by 10 percent or more from a previously recorded value; or radiographic changes indicative of pulmonary function.
Time Frame: Baseline up to Week 192
Population: ITT population included all participants who had at least 1 post-baseline efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Ataluren
Number analyzed (Participants) | 60
percentage of participants | 58.3

7. Secondary Outcome: Change From Baseline in 12-Lead Electrocardiogram (ECG) Parameters at Final Visit (Week 196)
Description: ECG parameters included RR duration, PR duration, QRS duration, QT duration, QTCB (Bazett's correction formula) duration, QTCF (Fridericia's correction formula) duration.
Time Frame: Baseline, Week 196
Population: As-treated population included all participants who received at least 1 dose of ataluren. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure. 'Number analyzed' signifies participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: miiliseconds
Arm/Group | Ataluren
Number analyzed (Participants) | 59
miiliseconds
  Baseline: RR duration | 828.17 (132.15)
  Change at Week 196: RR duration: number analyzed (Participants) | 55
  Change at Week 196: RR duration | -14.27 (115.62)
  Baseline: PR duration | 145.02 (19.29)
  Change at Week 196: PR duration: number analyzed (Participants) | 55
  Change at Week 196: PR duration | -2.69 (12.25)
  Baseline: QRS duration | 83.90 (8.00)
  Change at Week 196: QRS duration: number analyzed (Participants) | 55
  Change at Week 196: QRS duration | 0.33 (6.12)
  Baseline: QT duration | 370.71 (28.11)
  Change at Week 196: QT duration: number analyzed (Participants) | 55
  Change at Week 196: QT duration | -4.38 (25.63)
  Baseline: QTCB duration | 408.92 (22.05)
  Change at Week 196: QTCB duration: number analyzed (Participants) | 55
  Change at Week 196: QTCB duration | -0.71 (17.96)
  Baseline: QTCF duration | 395.47 (19.23)
  Change at Week 196: QTCF duration | -2.27 (17.13)

8. Secondary Outcome: Change From Baseline in Heart Rate at Final Visit (Week 196), as Assessed by 12-Lead ECG
Description: Heart rate was measured using 12-lead ECG.
Time Frame: Baseline, Week 196
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Ataluren
Number analyzed (Participants) | 59
beats/minute
  Baseline | 74.31 (12.06)
  Change at Week 196: number analyzed (Participants) | 55
  Change at Week 196 | 2.04 (10.11)

9. Secondary Outcome: Change From Baseline in Vital Signs at Final Visit (Week 196)
Description: Vital Signs included systolic blood pressure (SBP) and diastolic blood pressure (DBP).
Time Frame: Baseline, Week 196
Population: As-treated population included all participants who received at least 1 dose of ataluren. Here, 'Number analyzed' signifies participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Ataluren
Number analyzed (Participants) | 61
millimeters of mercury (mmHg)
  Baseline: SBP | 114.8 (9.10)
  Change at Week 196: SBP: number analyzed (Participants) | 59
  Change at Week 196: SBP | 0.6 (12.62)
  Baseline: DBP | 71.2 (8.93)
  Change at Week 196: DBP: number analyzed (Participants) | 59
  Change at Week 196: DBP | -0.3 (9.93)

10. Other Pre Specified Outcome: Change From Baseline in Percent Predicted Forced Vital Capacity (FVC) at the End of Treatment (Week 192), as Assessed by Spirometry
Description: FVC is the volume of air that can forcibly be blown out after full inspiration in the upright position. Percent of predicted FVC = (observed value)/(predicted value) * 100%. Change from baseline in percent predicted FVC at the end of treatment was reported.
Time Frame: Baseline, Week 192
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of predicted FVC
Arm/Group | Ataluren
Number analyzed (Participants) | 59
percentage of predicted FVC
  Baseline | 73.576 (14.6552)
  Change at Week 192: number analyzed (Participants) | 7
  Change at Week 192 | -2.286 (4.5722)

11. Other Pre Specified Outcome: Change From Baseline in Percent Predicted Forced Expiratory Flow Between 25% and 75% of Expiration (FEF25-75) at the End of Treatment (Week 192), as Assessed by Spirometry
Description: FEF25-75 is the forced expiratory flow between 25 and 75% of vital capacity.
Time Frame: Baseline, Week 192
Population: Due to change in planned analysis FEV25-75 was not calculated and summarized.
Arm/Group | Ataluren
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to end of study (Week 196)
Description: As-treated population included all participants who received at least 1 dose of ataluren.
Arm/Group | Ataluren
All-Cause Mortality (participants affected / at risk) | 1/61
Serious Adverse Events (participants affected / at risk) | 36/61
Other Adverse Events (participants affected / at risk) | 61/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren (N=61)
Appendicitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 27
Viral upper respiratory tract infection (Infections and infestations) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Distal ileal obstruction syndrome (Gastrointestinal disorders) | 1
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 3
Intestinal obstruction (Gastrointestinal disorders) | 1
Blood creatine increased (Investigations) | 1
Forced expiratory volume decreased (Investigations) | 2
Pulmonary function test decreased (Investigations) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Cystic fibrosis (Congenital, familial and genetic disorders) | 1
Gallbladder pain (Hepatobiliary disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren (N=61)
Gastroenteritis (Infections and infestations) | 5
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 50
Influenza (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 5
Oral candidiasis (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 9
Viral upper respiratory tract infection (Infections and infestations) | 22
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 8
Haemorrhoids (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4
Drug hypersensitivity (Immune system disorders) | 5
Headache (Nervous system disorders) | 5

LIMITATIONS AND CAVEATS:
Based on the results of study PTC124-GD-021-CF (NCT02139306) (did not achieve its primary or secondary endpoints), clinical development of ataluren in cystic fibrosis was discontinued and this ongoing open-label extension study was closed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT02107859/SAP_000.pdf
  • Study Protocol (2016-02-08): https://cdn.clinicaltrials.gov/large-docs/59/NCT02107859/Prot_001.pdf